CLINICAL TRIAL: NCT02159950
Title: A Phase II Randomized Open Label Study of Sipuleucel-T vs. Sipuleucel-T and Tasquinimod in Patients With Metastatic Castrate-Resistant Prostate Cancer (CRPC)
Brief Title: Sipuleucel-T With or Without Tasquinimod in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 250813; NCI-2014-01184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 250813 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2014-06-09; First posted 2014-06-10 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T; tasquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (sipuleucel-T) (Experimental): Patients receive sipuleucel-T IV over 60 minutes on day 4. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Sipuleucel-T
- Arm II (tasquinimod, sipuleucel-T) (Experimental): Patients receive tasquinimod PO QD beginning on day -14 and sipuleucel-T IV over 60 minutes on day 4. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients continue on tasquinimod treatment after day 42 until disease progression.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Sipuleucel-T; Drug: Tasquinimod

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Sipuleucel-T — Given IV
  Other Names: APC8015; APC8015 Vaccine; PA2024 (PAP/GM-CSF)-Loaded Dendritic Cell Vaccine; Provenge
Drug: Tasquinimod — Given PO
  Other Names: ABR-215050; TASQ
  Arms: Arm II (tasquinimod, sipuleucel-T)

SUMMARY:
This randomized phase II trial studies how well sipuleucel-T with or without tasquinimod works in treating patients with hormone-resistant prostate cancer that has spread to other parts of the body. Vaccines made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells. Tasquinimod may stop the growth of prostate cancer by blocking the growth of new blood vessels necessary for tumor growth. It is not yet known whether sipuleucel-T is more effective with or without tasquinimod in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether tasquinimod augments immune response to sipuleucel-T.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of sipuleucel-T and tasquinimod in patients with castration-resistant metastatic prostate cancer.

II. To obtain preliminary evidence of the clinical benefit of the combination of sipuleucel-T and tasquinimod; to include changes in prostate specific antigen (PSA) over time, and duration of progression-free survival/overall survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive sipuleucel-T intravenously (IV) over 60 minutes on day 4. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive tasquinimod orally (PO) once daily (QD) beginning on day -14 and sipuleucel-T IV over 60 minutes on day 4. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients continue on tasquinimod treatment after day 42 until disease progression.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic asymptomatic or minimally symptomatic castration-resistant prostate cancer (CRPC) patients who are eligible for sipuleucel-T
* Disease progression by PSA criteria (PSA Working Group Consensus Criteria Eligibility) and/or Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Life expectancy >= 6 months
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Hemoglobin >= 100 g/L (>= 10 g/dL)
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 x laboratory upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x laboratory upper limit of normal
* Creatinine =< 1.5 x laboratory upper limit of normal or calculated creatinine clearance of >= 50 mL/min (please use institutional formula)
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5
* Urine protein < 1+; if >= 1+, 24 hour urine protein should be obtained and should be < 1000 mg
* Central nervous system (CNS): no recent history (within 6 month) of cerebrovascular accident, transient ischemic attacks, central nervous system or brain metastases
* Ability to understand and the willingness to sign a written informed consent document
* Patient verbalizes the ability to swallow and retain oral medication
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have received systemic steroids within 4 weeks prior to starting study treatment
* Patients who have received prior immunotherapies
* History of therapy for an autoimmune disorder
* Patients receiving any other investigational agents
* Any medical condition that would preclude adequate evaluation of the safety and toxicity of the study combination
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Association class II, III, or IV), angina pectoris requiring nitrate therapy, recent myocardial infarction (less than the last 6 months), cardiac arrhythmia, history of cerebrovascular accident (CVA) within 6 months; no uncontrolled hypertension (defined as blood pressure of > 160/90 mmHg) on medication or, history of peripheral vascular disease
* Ongoing treatment with warfarin unless the international normalized ratio (INR) is well controlled and below 4
* History of psychiatric illness or social situations that would limit compliance with study requirements
* History of pancreatitis
* Human immunodeficiency virus (HIV)-positive patients receiving combination antiretroviral therapy are ineligible
* Systemic exposure to ketoconazole or other strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) isoenzyme inhibitors or inducers within 14 days prior to the start of study treatment; systemic exposure to aminodarone is not allowed within 1 year prior to the start of study treatment
* Ongoing treatment with sensitive cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) substrate or CYP1A2 substrate with narrow therapeutic range at the start of study treatment
* Ongoing treatment with CYP3A4 substrate with narrow therapeutic range at the start of study treatment
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of therapy
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T) | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 75.4 (.70) | 75.4 (.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Immune Response Assessed by IFN-g ELISPOT Specific for PA2024
Time Frame: Baseline up to 50 weeks
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in PSA Response
Description: PSA doubling time, PSA slope
Time Frame: Baseline to up to 3 years
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Duration of PSA Response
Time Frame: Up to 3 years
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Frequency of Toxicities Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4
Description: The frequency of participants with toxicities will be tabulated by grade across all dose levels and courses.
Time Frame: Up to 3 years
Population: All treated and eligible patients.
Measure: Number; unit: participants
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 2
participants
  Grade 1 |  | 1
  Grade 4 |  | 1

5. Secondary Outcome: Immune Response
Time Frame: Week 6
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Immune Response
Time Frame: Week 10
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Immune Response
Time Frame: Week 26
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Immune Response
Time Frame: Week 50
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Immune Response (Arm 2 Only)
Time Frame: Week 0
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Objective Response Rates (Partial or Complete)
Time Frame: Up to 3 years
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Overall Survival
Time Frame: Up to 3 years
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Progression-free Survival
Time Frame: Up to 3 years
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Time to PSA Progression
Time Frame: Up to 3 years
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Effects of Tasquinimod on the Inhibition of Immune Cells
Time Frame: Up to week 50
Population: Due a Lack of funding data was not collected and no patients were analyzed.
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Sipuleucel-T) | Arm II (Tasquinimod, Sipuleucel-T)
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/2
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sipuleucel-T) (N=0) | Arm II (Tasquinimod, Sipuleucel-T) (N=2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sipuleucel-T) (N=0) | Arm II (Tasquinimod, Sipuleucel-T) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (23)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (30)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (10)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (57)
Fatigue (General disorders) | 0 (0) | 2 (27)
Malaise (General disorders) | 0 (0) | 1 (18)
Weight decreased (Investigations) | 0 (0) | 1 (8)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (13)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (24)

LIMITATIONS AND CAVEATS:
Due to the study's early closure, as a result of lack of funding, target accrual was not reached and no statistical inference of the primary and secondary aims were carried forth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes